CLINICAL TRIAL: NCT06826027
Title: TAV-in-SAV in Japanese Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Osaka University (Other)
Collaborators: Medtronics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TAV-in-SAV in Japan
Record Dates: First submitted 2025-01-11; First posted 2025-02-13 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-02

CONDITIONS: Valve-in-valve Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- TAV-in-SAV

SUMMARY:
Background In 2018, transcatheter aortic valve in surgical aortic valve (TAV-in-SAV) in high risk patients was approved for the treatment of bioprosthetic valve dysfunction due to aging, for which valve replacement had been selected. It has been reported that early and mid-term results of TAV-in-SAV differ depending on the sizes of the original surgical bioprosthetic valves. Especially, the prognoses of TAV-in-SAV in patients with surgical bioprosthetic valves of ≤21 mm in size are reported to be poor in the United States and Europe. Bioprosthetic valves of ≥21 mm in size are thus tended to be used also in Japan after the annular was enlarged in the initial surgery as needed. The patient group in the above-mentioned report, however, consisted of larger patients (with the mean body surface area of 1.85 m2). It has therefore been unknown whether the above report applies to smaller patients in Japan. Furthermore, in terms of the surgical results for valvular disease, not only short-term results, but also repeat surgery avoidance rate, as well as medium- and long-term results, including the occurrence rate of complications related to artificial valves, are important factors, but the characteristic of this disease, the number of cases at each facility is not that large, so there have been no comprehensive reports of TAV-in-SAV in Japan. Accordingly, the investigators will investigate TAV-in-SAV performed at Osaka University as well as multiple centers in Japan to: understand the facts; assess the appropriateness of the evaluation of the above-mentioned paper; and examine early and mid-term treatment results of TAV-in-SAV in patients with narrow bioprosthetic valves, which are specific to Japanese patients. The investigators also plan to study early and mid-term treatment results of TAV-in-SAV using a self-expanding valve because self-expanding valves generally produce favorable hemodynamics in narrow bioprosthetic valves.

Study Objectives i. To study early and mid-term results of transcatheter aortic valve implantation in patients with aortic bioprosthetic valve dysfunction (hereinafter referred to as TAV-in-SAV).

ii. To compare clinical results, including hemodynamics, of TAV-in-SAV between small aortic bioprosthetic valves (19 or 21 mm in size) and aortic bioprosthetic valves of other sizes.

iii. To compare clinical results, including hemodynamics, of TAV-in-SAV between a self-expanding valve and a balloon-expandable valve.

Study Methods i. Study design A multicenter, retrospective, observational study using existing data. ii. Endpoints

Study endpoints are as follows:

Primary endpoint: Death during the observation period The mortality among all patients registered in this study will be estimated with the Kaplan-Meier method.

Secondary endpoints: Analyses of major cardiac and cerebral events (MACCE) and factors associated with death. The rate of freedom from MACCE among all patients registered in this study will be estimated with the Kaplan-Meier method. Factors associated with death will be explored using a Cox proportional hazards model.

Hemodynamics and events including death and MACCE will also be compared between aortic bioprosthetic valves of 19 or 21 mm in size and those of other sizes.

In addition, hemodynamics and events including death and MACCE will be compared between a self-expanding valve (Evolut) and a balloon-expandable valve (SAPIEN) using propensity-matching analyses.

ELIGIBILITY:
Inclusion Criteria:

This study will include patients who underwent TAV-in-SAV at the Osaka University Hospital or any of the following study centers between January 1, 2013 and March 31, 2023.

Exclusion Criteria:

Study subjects who or whose legally accepted representatives refuse to participate in or to continue to be in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will include patients who underwent TAV-in-SAV at the Osaka University Hospital or any of the following study centers between January 1, 2013 and March 31, 2023.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2024-08-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Death during the observation period | through study completion, an average of 2 year

SECONDARY OUTCOMES:
freedom from MACCE | through study completion, an average of 2 year

CONTACTS AND LOCATIONS:
Locations (10):
- Japan (10):
  - Tokyo Bay Urayasu Ichikawa Medical Center, Urayasu, Chiba
  - Kyusyu University, Fukuoka, Fukuoka
  - Kurume University, Kurume, Kurume
  - The Skakibara Heart Institute of Okayama, Okayama, Okayama-ken
  - Osaka International Medical and Science Center, Osaka, Osaka
  - Osaka University, Suita, Osaka
  - Saga University, Saga, Saga-ken
  - Dokkyo Medical University Saitama Medical Center, Koshigaya, Saitama
  - Tokyo Women's Medical University, Shinjuku, Tokyo
  - Tottori University, Yonago, Tottori

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dvir D, Webb JG, Bleiziffer S, Pasic M, Waksman R, Kodali S, Barbanti M, Latib A, Schaefer U, Rodes-Cabau J, Treede H, Piazza N, Hildick-Smith D, Himbert D, Walther T, Hengstenberg C, Nissen H, Bekeredjian R, Presbitero P, Ferrari E, Segev A, de Weger A, Windecker S, Moat NE, Napodano M, Wilbring M, Cerillo AG, Brecker S, Tchetche D, Lefevre T, De Marco F, Fiorina C, Petronio AS, Teles RC, Testa L, Laborde JC, Leon MB, Kornowski R; Valve-in-Valve International Data Registry Investigators. Transcatheter aortic valve implantation in failed bioprosthetic surgical valves. JAMA. 2014 Jul;312(2):162-70. doi: 10.1001/jama.2014.7246. PMID 25005653